CLINICAL TRIAL: NCT06213246
Title: Effect of Surgery and Sleep Hygiene Strategies on Strength, Sleep Parameters, and Cognitive Performance in Orthopedic Surgeons
Brief Title: Sleep and Performance in Surgeons
Acronym: Sleep&Surgeon
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Sleep&Surgeons (L4157)
Record Dates: First submitted 2023-12-22; First posted 2024-01-19 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Sleep
Keywords: surgery; sleep; surgeon; strength; cognitive performance

STUDY DESIGN:
Intervention Model Description: The study is monocentric, prospective, and observational.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sleep Hygiene Strategies (SHS) (Experimental): In Week 3, the study participants will implement sleep hygiene strategies. Specifically, these sleep hygiene strategies will be applied for all seven days of Week 3 and will involve the guidelines recommended by the National Sleep Foundation.
  Interventions: Behavioral: Sleep Hygiene Strategies

INTERVENTIONS:
Behavioral: Sleep Hygiene Strategies — The sleep hygiene strategies will be applied for all seven days of Week 3 and will involve the following guidelines recommended by the National Sleep Foundation
  * Maintain a consistent wake-up and bedtime schedule during workdays.
  * Do not delay/advance excessively (no more than 2 hours) the wake-up and bedtime - schedule during weekends.
  * Keep the bedroom temperature below 22°C.
  * Avoid sources of light and noise in the bedroom.
  * Use the bed only for sleeping, avoiding other activities before bedtime.
  * Avoid daytime naps during workdays.
  * Refrain from using electronic devices (PC, laptop, cellphone, television) at least 30 minutes before bedtime.
  * Expose yourself to natural light in the morning and reduce artificial lights in the evening.
  * Avoid consuming alcoholic beverages and caffeine in the afternoon.
  * Have a moderately sized dinner at least 3 hours before bedtime.

SUMMARY:
The primary aim of this study is to assess the changes in strength expression resulting from the performance of a surgical operation among orthopedic surgeons at the IRCCS Galeazzi-Sant'Ambrogio Hospital. To achieve this goal, the assessment of strength expression will be conducted using handgrip measurements before (pre) and after (post) the surgical operation. Additionally, both pre- and post-surgery, there will also be evaluations of changes in actigraphic sleep parameters, salivary cortisol levels, cognitive performance, and subjective perception levels of effort and drowsiness.

Te second aim is to assess differences in strength expression, cognitive performance, salivary cortisol levels, perceived effort, and drowsiness levels among surgeons in response to sleep hygiene strategies (week 2 vs week 3).

DETAILED DESCRIPTION:
Currently, there are few scientific studies that have assessed the relationship between sleep quality, strength expression, and cognitive performance among orthopedic surgeons. Furthermore, no previous study has ever evaluated the effect of a behavioral sleep hygiene strategy on actigraphic sleep parameters in orthopedic surgeons.

Therefore, the primary aim of the study is to assess the changes in strength expression resulting from the performance of a surgical operation among orthopedic surgeons at the IRCCS Galeazzi-Sant'Ambrogio Hospital. To achieve this goal, the assessment of strength expression will be conducted using handgrip measurements before (pre) and after (post) the surgical operation. Additionally, both pre- and post-surgery, there will also be evaluations of changes on lower limbs strength (maximal isometric strength of extensors of knee by digital dynamometer), salivary cortisol levels, cognitive performance (Stroop test and Bomb Risk Elicitation Task), and subjective perception levels of effort and drowsiness (Borg CR-10 and Karolinska Sleepiness Scale).

Te second aim is to assess differences in strength expression, cognitive performance, salivary cortisol levels, perceived effort, and drowsiness levels among surgeons in response to sleep hygiene strategies (control week vs Sleep hygiene strategies week).

The study involves 3 weeks of assessment (Week 1, 2, and 3), not necessarily consecutive.

Assessments within Week 1:

- Sleep monitoring using actigraphy and a sleep diary for the entire week, along with completing the Morningness-Eveningness Questionnaire and Pittsburgh Sleep Quality Index.

Assessments within Week 2 and Week 3:

* Sleep monitoring using actigraphy and a sleep diary for the entire week.
* Pre and post-surgical operation evaluations:

  * Measurement of strength using dynamometers.
  * Cognitive assessment using Stroop test and Bomb Risk Elicitation Task.
  * Evaluation of salivary cortisol levels using "Salivette".
  * Assessment of perceived exertion using the Borg CR10 scale.
  * Evaluation of drowsiness levels using the Karolinska Sleepiness Scale.

Note: In Week 3, sleep hygiene strategies will be implemented.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, of any ethnicity;
* Age between 23 and 70 years old;
* Cognitively intact;
* Orthopedic surgeons or medical residents specializing in Orthopedics.
* Signature and acceptance of informed consent to collaborate in all procedures necessary for the study.

Exclusion Criteria:

* Individuals younger than 23 years old or older than 70 years old;
* Any clinical condition that prevents the subject from participating in operating room activities (e.g., muscle injury, COVID-19 positivity, feverish or flu-like states, etc.).
* Non-participation, for any reason, in surgical activities in daily clinical practice.
* Clinically diagnosed sleep disorders.
* Women who have been pregnant or breastfeeding within 12 months before signing the informed consent or during the recruitment and observation period. [self-declaration]
* Non-acceptance of the informed consent.
* Physical impossibility to undergo the evaluations required by the study using the devices specified in the protocol.

Ages: 23 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2023-10-23 (Actual); Primary Completion 2024-12-23 (Estimated); Study Completion 2024-12-23 (Estimated)

PRIMARY OUTCOMES:
Handgrip Test | The handgrip test is conducted on the seventh day of both Week 2 and Week 3, taking approximately 4 minutes to complete. The test is performed both before and after the surgery.
  Handgrip is a measure of the maximal isometric force that a hand can squeeze, and it is widely used because very easy and inexpensive. The handgrip strength is performed three-times for each hand alternatively, starting with the dominant hand, using a digital dynamometer to the nearest 0.1kg. Participants perform the test in a sitting position with the shoulder adducted, elbow flexed at 90-degree angle, forearm in neutral position. Participants rest 30 seconds among each repetition. The peak of the three repetitions is calculated and use for statistical analysis.

SECONDARY OUTCOMES:
Lower limbs isometric strength | The maximal isometric strength test of extensors of knee is conducted on the seventh day of both Week 2 and Week 3, taking approximately 5 minutes to complete. The test is performed both before and after the surgery.
  Maximal isometric strength of extensors of knee is measured, for both lower limbs alternatively, using a digital dynamometer with subjects in a sitting position and the knee placed at 90° flexion. A resting period of 30-seconds is given after each repetition. The peak of the three repetitions is calculated and used for statistical analysis.
Sleep monitoring | Seven days for each timepoint period (week 1, week 2 and week 3. 21 days in total)
  Sleep parameters are objectively monitored by actigraphy. Also, participants complete a validated daily sleep diary to record bedtime, wake-up time, the number and duration of nocturnal awakenings, daytime napping, and subjective sleep quality. Data derive both from the sleep device and sleep diaries are used to determine the quantity and quality of sleep that participants obtain (Total sleep time; Sleep efficiency; Immobility time; Moving time; Fragmentation index; Wake after sleep onset; Subjective quality of sleep; Subjective sleepiness; Subjective tiredness). Sleep is monitored for seven consecutive days for each timepoint period (week 1, week 2 and week 3).
Stroop Test | The Stroop test is conducted on the seventh day of both Week 2 and Week 3, taking approximately 2 minutes to complete. The test is performed both before and after the surgery.
  The Stroop test is a psychological assessment that evaluates cognitive processing speed and selective attention. The Stroop test involves presenting words in different colors and asking participants to name the color of the ink used to print the word.
Bomb Risk Elicitation Task | The Bomb Risk Elicitation Task is conducted on the seventh day of both Week 2 and Week 3, taking approximately 2 minutes to complete. The test is performed both before and after the surgery.
  The Bomb Risk Elicitation Task is a behavioral experiment designed to measure risk preferences under uncertainty. The task involves decision-making in a context where participants face varying levels of risk and potential gains or losses.
Salivary cortisol | The assessment of salivary cortisol using "Salivette" is conducted on the seventh day of both Week 2 and Week 3, taking approximately 3 minutes to complete. The assessment is performed both before and after the surgery.
  Assessment of salivary cortisol levels using Salivette tubes (Sarsted, Germany)
Borg CR-10 | The Borg CR-10 evaluation is conducted on the seventh day of both Week 2 and Week 3, taking approximately 1 minute to complete. The assessment is performed both before and after the surgery.
  Borg CR-10 is a tool used to measure subjective perception of exertion during physical activity. This scale assesses an individual's subjective perception of effort or exertion during exercise, ranging from 0 (no exertion at all) to 10 (maximal exertion).
Karolinska Sleepiness Scale | The Karolinska Sleepiness Scale evaluation is conducted on the seventh day of both Week 2 and Week 3, taking approximately 1 minute to complete. The assessment is performed both before and after the surgery.
  The Karolinska Sleepiness Scale is a subjective self-assessment tool used to measure a person's level of sleepiness or alertness at a particular moment in time. This scale helps individuals rate their perceived sleepiness on a scale from 1 (Very alert) to 9 (Extremely sleepy, can't stay awake).
Pittsburgh Sleep Quality Index | The Pittsburgh Sleep Quality Index evaluation is conducted at the end of Week 1, and taking approximately 4 minute to complete.
  The Pittsburgh Sleep Quality Index is a widely used self-report questionnaire that assesses an individual's sleep quality over a one-month time interval. It evaluates various aspects of sleep, including duration, latency, habitual sleep efficiency, disturbances, use of sleep medications, and daytime dysfunction. The global score ranging from 0 to 21, where higher scores indicate poorer sleep quality.
Morningness-Eveningness Questionnaire | The Morningness-Eveningness Questionnaire is conducted at the end of Week 1, and taking approximately 4 minute to complete.
  The Morningness-Eveningness Questionnaire (MEQ) is a self-report questionnaire designed to assess an individual's chronotype, which refers to their preference for being active and alert during certain parts of the day. Based on the responses, individuals are scored on a scale (range from 16 to 86) that categorizes them into different chronotypes:
  * Morning types (score: 59-86)
  * Intermediate types (score: 42-58)
  * Evening types (score: 16-41)

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Ospedale Galeazzi-Sant'Ambrogio, Milan, Italy